CLINICAL TRIAL: NCT06275724
Title: Specified Drug-use Survey of Leqvio for s.c. Injection (Familial Hypercholesterolaemia or Hypercholesterolaemia, CKJX839A11401)
Brief Title: Specified Drug-use Survey of Leqvio for s.c. Injection.
Status: Active, not recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A11401
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Familial Hypercholesterolaemia; Hypercholesterolaemia
Keywords: familial hypercholesterolaemia; hypercholesterolaemia; FH; HoFH; Leqvio; inclisiran sodium
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Homozygous Familial Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- inclisiran: Patients prescribed with inclisiran
  Interventions: Other: inclisiran

INTERVENTIONS:
Other: inclisiran — Prospective observational study. There is no treatment allocation. Patients prescribed with inclisiran are eligible to enroll into this study.

SUMMARY:
The objective of this study is to evaluate the long-term safety of Leqvio in patients with familial hypercholesterolaemia or hypercholesterolaemia in post-marketing clinical practice

DETAILED DESCRIPTION:
Uncontrolled, central registration system, multicenter, special drug use-results surveillance.

This is a prospective, open-label, multicenter, single-arm observational study (non-interventional study: NIS) conducted only in Japan.

The survey will include patients with familial hypercholesterolaemia or hypercholesterolaemia who have received treatment with Leqvio. Patients who discontinued treatment with Leqvio before completing the 24-month observation period will be followed for safety until the date of the last dose of Leqvio plus 180 days or until 24 months after the first dose of Leqvio, whichever comes earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provided written informed consent to participate in this survey prior to the start of treatment with Leqvio.
* Patients who received treatment with Leqvio as per the package insert.

Exclusion Criteria:

* Patients who received treatment with a formulation containing the same ingredients as Leqvio in the past.
* Patients participating in other interventional studies at the time of informed consent.
* Patients planning to participate in other interventional studies during this survey.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with inclisiran
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 24 months
  To evaluate the long-term safety profile of Leqvio
Numbers of patients with serious adverse events, adverse events by severity, and adverse drug reactions | Up to 24 months
  To evaluate the long-term safety profile of Leqvio

SECONDARY OUTCOMES:
Number of patients with adverse events leading to discontinuation of treatment with the product | Up to 24 months
  To evaluate the tolerability of Leqvio
Percent change from baseline in LDL-C levels | Month 24
  To evaluate the efficacy of Leqvio based on LDL-C levels

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (89):
- Japan (89):
  - Novartis Investigative Site, Handa, Aichi-ken
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Komaki, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Tsushima, Aichi-ken
  - Novartis Investigative Site, Asahi, Chiba
  - Novartis Investigative Site, Inzai, Chiba
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukui-shi, Fukui
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Kōriyama, Fukushima
  - Novartis Investigative Site, Shirakawa, Fukushima
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Ono, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Kamisu, Ibaraki
  - Novartis Investigative Site, Koga, Ibaraki
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Moriya, Ibaraki
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Fujisawa, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Yatsushiro, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Kyōtanabe, Kyoto
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Ikoma, Nara
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Tenri, Nara
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Urasoe, Okinawa
  - Novartis Investigative Site, Uruma, Okinawa
  - Novartis Investigative Site, Izumisano, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Toyonaka, Osaka
  - Novartis Investigative Site, Asaka, Saitama
  - Novartis Investigative Site, Gyōda, Saitama
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Kitamoto, Saitama
  - Novartis Investigative Site, Sōka, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Nagahama, Shiga
  - Novartis Investigative Site, Izunokuni, Shizuoka
  - Novartis Investigative Site, Mooka, Tochigi
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Minato, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Shinjuku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Sumida City, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
  - Novartis Investigative Site, Takaoka, Toyama
  - Novartis Investigative Site, Hashimoto, Wakayama
  - Novartis Investigative Site, Sakata, Yamagata
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Himeji
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Nara
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka

IPD SHARING:
Plan to Share IPD: No